CLINICAL TRIAL: NCT02168205
Title: Hase I Open-Label Two-Part Study To Evaluate The Effect Of Food and Of CYP1A2 Induction On Pomalidomide (CC-4047) Pharmacokinetics in Healthy Subjects
Brief Title: Food Effect and CYP1A2 Induction Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CC-4047-CP-011
Expanded Access: NCT03723096 (No longer available)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteer; Pharmacokinetics; Pomalyst; Pomalidomide; Food effect; smoker
MeSH Terms: interventions — pomalidomide; Caffeine; Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4 mg Pomalidomide - Fed (Experimental): On Day 1, participants will receive a single oral dose of 4 mg pomalidomide under fed conditions.
  Interventions: Drug: Pomalidomide
- 4 mg Pomalidomide - Fasted (Experimental): On Day 1, participants will receive a single oral dose of 4 mg pomalidomide under fasted conditions
  Interventions: Drug: Pomalidomide
- 4 mg Pomalidomide + caffeine - Non-smoking (Experimental): Participants will remain in the clinical site for a total of 10 days. They will receive orally a 200-mg caffeine capsule on Day 6, and on Day 8, participants will receive a single oral dose of 4 mg pomalidomide.
  Interventions: Drug: Pomalidomide; Other: Caffeine
- 4 mg Pomalidomide + caffeine - Smoking (Experimental): Participants will be required to smoke approximately 20 cigarettes a day for 10 days. They will receive orally a 200-mg caffeine capsule on Day 6, and on Day 8, participants will receive a single oral dose of 4 mg pomalidomide.
  Interventions: Drug: Pomalidomide; Other: Caffeine; Other: Tobacco

INTERVENTIONS:
Drug: Pomalidomide — Capsules
Other: Caffeine — Capsules
  Arms: 4 mg Pomalidomide + caffeine - Non-smoking; 4 mg Pomalidomide + caffeine - Smoking
Other: Tobacco — Cigarettes
  Arms: 4 mg Pomalidomide + caffeine - Smoking

SUMMARY:
This study will evaluate the effect of food and smoking on healthy older subjects taking pomalidomide.

DETAILED DESCRIPTION:
This study will be conducted in two parts. Parts 1 and 2 may be conducted in parallel and subjects are only allowed to participate in one part.

In Part 1, subjects will be randomly assigned to receive a single oral dose of 4 mg pomalidomide on Day 1 under fed (standard high fat breakfast) or fasted conditions. After a washout period of at least 3 and no more than 7 days, subjects will receive a single oral dose of 4 mg pomalidomide under the opposite condition to what they received in the first period.

In Part 2, healthy male smoker subjects must smoke approximately 20 cigarettes per day for a total of 10 days. Non-smokers will neither smoke nor be in the presence of smokers. All subjects will receive orally a 200-mg caffeine capsule on Day 6, and on Day 8, subjects will receive a single oral dose of 4 mg pomalidomide.

For both Parts 1 and 2, serial blood samples will be collected for determination of plasma pomalidomide concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: 1.Must understand and voluntarily sign a written Informed Consent prior to any study-related procedures being performed.

  2.Must be able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.

  3.Must be male or postmenopausal* women of any race between ≥61 to ≤85 years of age (inclusive) at the time of signing the Informed Consent, and in good health as determined by a physical exam, clinical laboratory safety test results, vital signs, and 12 lead Electrocardiogram.

  * =Naturally postmenopausal for at least 24 consecutive months (ie, who has not had menses at any time in the preceding 24 consecutive months) 4.Subjects must be a non smoker. 5.Clinical laboratory tests must be within normal limits or acceptable to the Principal Investigator (PI).

  6.Must have a normal or clinically acceptable 12-lead Electrocardiogram. 7.Must be afebrile (febrile is defined as ≥ 38.0ºC or 100.4 Fahrenheit), with supine systolic blood pressure (BP): 90 to 150 mmHg, supine diastolic blood pressure: 60 to 95 mmHg, and pulse rate: 40 to 110 bpm and controlled on medications if they are indicated (especially for blood pressure).
  1. If a subject has a diagnosis of hypertension, the range for BP and pulse rate will be the one that is considered well controlled on medication.

     8.Must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female that can get pregnant while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.

     * = True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Period abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception 9.Must agree to refrain from donating sperm or semen while participating in this study and for at least 28 days following the last dose of study drug.

     10.Must agree to refrain from donating blood or plasma (other than for this study) while participating in this study and for at least 28 days following the last dose of study drug.

     11.Must agree to comply with the conditions described in the counseling document (part of the pomalidomide Pregnancy Prevention Risk Management Plan.

     Part 2
     1. Must understand and voluntarily sign a written informed consent prior to any study-related procedures being performed.
     2. Must be able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
     3. Must be male of any race between 40 to 80 years of age (inclusive) at the time of signing the Informed Consent, and in good health as determined by a physical exam, clinical laboratory safety test results, vital signs, and 12 lead electrocardiogram.
     4. Cohort A subjects (smokers) must have a history of smoking for >5 years and currently smoke ≥1 pack (20-25) cigarettes per day; and urine cotinine level at screening and baseline (Day -1) indicate subject is heavy smoker.
     5. Cohort B subjects (non-smokers) must have not smoked for >5 years (Cohort B).
     6. Clinical laboratory tests must be within normal limits or acceptable to the Principal Investigator.
     7. Must have a normal or clinically acceptable 12-lead Electrocardiogram, with a QTcF value ≤ 450 msec.
     8. Must be afebrile (febrile is defined as ≥ 38.0ºC or 100.4 Fahrenheit), with supine systolic blood pressure (BP): 90 to 150 mmHg, supine diastolic blood pressure: 60 to 95 mmHg, and pulse rate: 40 to 110 bpm and controlled on medications if they are indicated (especially for blood pressure).
     9. Must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female that can get pregnant while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.
     10. Must agree to refrain from donating sperm or semen while participating in this study and for at least 28 days following the last dose of study drug.
     11. Must agree to refrain from donating blood or plasma (other than for this study) while participating in this study and for at least 28 days following the last dose of study drug.
     12. Must agree to comply with the conditions described in the counseling document (part of the pomalidomide Pregnancy Prevention Risk Management Plan.

     Exclusion Criteria:
* Both Parts:

  1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, known hypersensitivity to a member of the class of drugs that can modulate the immune system, or other major disorders.

     1. Subjects with well-controlled hypertension, hyperlipidemia, gout, asthma/chronic obstructive pulmonary disease, hypothyroidism and other common age-related disorders, requiring treatment and being well-controlled on concomitant prescription medication(s) will be eligible for inclusion in the study.
     2. Subjects with diabetes, significant gastrointestinal diseases or hematologic disorders should not be included in the study.
  2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
  3. Used any prescribed systemic or topical medication within 30 days of the first dose administration, unless these medications are chronically administered and Sponsor agreement is obtained.
  4. Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, unless these medications are chronically administered and Sponsor agreement is obtained.
  5. Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion, e.g., bariatric procedure.
  6. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
  7. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs.
  8. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or positive alcohol screen.
  9. Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen, or hepatitis C antibody, or have a positive result to the test for Human Immunodeficiency Virus antibodies at Screening.
  10. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
  11. Received vaccination (excluding seasonal flu vaccination) within 90 days of the study drug administration.
  12. Subjects who are part of the staff personnel or family members of the investigational study staff.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2014-09-19 (Actual); Study Completion 2014-09-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | Up to 8 days for Part 1; up to 10 days for Part 2
  Maximum observed concentration in plasma
Pharmacokinetics - Tmax | Up to 8 days for Part 1; up to 10 days for Part 2
  Time to maximum observed concentration in plasma
Pharmacokinetics - AUC | Up to 8 days for Part 1; up to 10 days for Part 2
  Area under the plasma concentration-time curve
Pharmacokinetics - T1/2 | Up to 8 days for Part 1; up to 10 days for Part 2
  Terminal half-life
Pharmacokinetics - Vz/f | Up to 8 days for Part 1; up to 10 days for Part 2
  Apparent volume of distribution
Pharmacokinetics - CL/F | Up to 8 days for Part 1; up to 10 days for Part 2
  Apparent total body clearance

SECONDARY OUTCOMES:
Adverse events | Approximately 1 month
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

REFERENCES:
- See also: Related Info — http://us.testwiththebest.com